CLINICAL TRIAL: NCT00394745
Title: A 12 Week Treatment, Open-label, Multicenter Study to Investigate the Efficacy and Safety of Valsartan 160-320 mg With Regard to Effects on Lipid Subfractions in Hypertensive Patients With Metabolic Syndrome
Brief Title: Effect of Valsartan on Lipid Subfractions in Hypertensive Patients With Metabolic Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVAL489ADE25
Record Dates: First submitted 2006-10-31; First posted 2006-11-01 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Hypertension; Metabolic Syndrome
Keywords: Hypertension, Metabolic Syndrome, lipid subfractions
MeSH Terms: conditions — Hypertension; Metabolic Syndrome | interventions — Valsartan

INTERVENTIONS:
Drug: Valsartan

SUMMARY:
The purpose of this study is to evaluate potential effects of valsartan on lipid subfractions and other parameters in lipid metabolism in patients with essential hypertension and metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients >= 18 years of age at Visit 1
* Hypertension (systolic blood pressure >= 140 mmHg and < 170 mmHg and/or diastolic blood pressure >= 90 mmHg and < 105 mmHg
* Elevated triglycerides
* Metabolic syndrome as defined by Adult Treatment Panel III criteria

Exclusion Criteria:

* MSSBP >= 170 mmHg and/or MSDBP >= 105 mmHg at any time between Visit 1 and Visit 2
* Diabetes mellitus
* Patients treated with lipid lowering drugs in the last 6 weeks prior to Visit 1
* A history of cardiovascular disease, including angina pectoris, myocardial infarction, coronary artery bypass graft, percutaneous transluminal coronary angioplasty, transient ischemic attack, stroke, and peripheral artery disease, heart failure NYHA II - IV Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2005-11; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of valsartan 320 mg on small, dense low density lipoprotein (LDL) subfractions in hypertensive patients with metabolic syndrome.

SECONDARY OUTCOMES:
To evaluate the effect of valsartan 320 mg on further lipid subfractions and enzymes related to the lipoprotein metabolism.
To evaluate the effect of valsartan 160-320 mg on blood pressure and pulse rate.
To assess the safety and tolerability of valsartan 160-320mg.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis + 41 61 324 1111 Basel, Study Director — Novartis Basel+ 41 61 324 1111
Locations (2):
- Investigative Centers, Germany
- Novartis, Basel, Switzerland